CLINICAL TRIAL: NCT05301673
Title: ADHD Remote Technology Study of Cardiometabolic Risk Factors and Medication Adherence ('ART-CARMA')
Brief Title: ADHD Remote Technology Study of Cardiometabolic Risk Factors and Medication Adherence
Acronym: ART-CARMA
Status: Active, not recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Barnet, Enfield and Haringey Mental Health NHS Trust (Other Government); Hospital Universitari Vall d'Hebron Research Institute (Other); Empatica, Inc. (Industry); Örebro University, Sweden (Other); Concentris research management gmbh (Unknown); Attention Deficit Disorder Information and Support Service (Unknown); The European Association for the Study of Obesity (Unknown); Northumberland, Tyne and Wear NHS Foundation Trust (Other); Tees, Esk and Wear Valleys NHS Foundation Trust (Unknown); South West London and St George's Mental Health NHS Trust (Other); East London NHS Foundation Trust (Other Government); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 304278
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Cardiovascular Diseases; Medication Adherence
Keywords: ADHD; attention-deficit/hyperactivity disorder; remote measurement technology; mHealth; cardiovascular disease; medication adherence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults with ADHD
- Partner, family member or close friend of the individuals with ADHD

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a common psychiatric disorder, with a prevalence among adults of 2.5%. The disorder is diagnosed based on impairing levels of inattentive, hyperactive and impulsive behaviours. Most adults with ADHD present with additional mental health problems. Adults with ADHD have an increased risk to develop so-called cardiometabolic illnesses, such as type-2 diabetes, obesity and cardiovascular disease (e.g., heart failure). However, detailed knowledge about the screening, diagnosis and management of adults with ADHD and co-occurring cardiometabolic illnesses is lacking. The purpose of ART-CARMA is to (1) obtain real-world data from adults with ADHD daily life on the extent to which ADHD medication treatment and physical activity, individually and jointly, may influence cardiometabolic risks in adults with ADHD, and (2) obtain real-world data of patterns of taking ADHD medication and reasons for not taking medication, over a remote monitoring period of 12 months.

ART-CARMA benefits from the ADHD Remote Technology ('ART') assessment and monitoring system for adults with ADHD (developed by Kuntsi, Dobson, et al.), and the RADAR-base mobile-health platform to which it is linked (developed by Dobson et al; http://www.radar-base.org). ART consists of both active (e.g., questionnaires) and passive (smartphone and a wearable device) monitoring. ART-CARMA will use remote measurement technology (RMT) in adults with ADHD to carry out unobtrusive, real-time data collection over a continuous period of 12 months. By recruiting 300 adults from adult ADHD clinic waiting lists (and a partner/family member/close friend for each of them) and monitoring them remotely, we will obtain objectively measured data relevant to cardiometabolic risk profiles from their daily lives. By targeting the period before starting any ADHD medication through to starting treatment and the subsequent period, up to 12 months in total, we obtain real-time data on multiple parameters, including side effects, that can inform the personalisation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-5 ADHD
* Aged 18-60
* Able to give informed consent for participation
* Fluent in English
* Willing and able to complete self-reported assessments via smartphone
* Willing to use either their own compatible Android phone or a study Android phone as their only smartphone during the data collection period
* Willing to wear the wearable device (EmbracePlus) during the data collection period
* Not on ADHD medication at the time of recruitment

Exclusion Criteria:

* Psychosis, currently experiencing a major depressive episode, mania, drug dependence in the last six months, or a major neurological disorder
* Recent contact with psychiatric acute care (admission, crisis team or liaison team (A&E)) in the last six months
* Any other major medical disease which might impact upon the patient's ability to participate in normal daily activities (e.g., due to hospitalisations)
* Pregnancy
* IQ < 70
* Does not start ADHD medication following ADHD diagnosis (either due to personal choice or psychiatrist deciding not to prescribe ADHD medication)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: There are two data collection sites. The KCL site will recruit 150 participants from adult ADHD clinics. The VHIR site will recruit 150 participants from their adult ADHD clinic.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | Continuously across a 12-month time period
  EmbracePlus wearable device
Change in blood pressure | Baseline and every 4 weeks up to month 12
  Blood pressure will be measured by participant
Change in weight | Baseline and every 4 weeks up to month 12
  Weight (in kg) will be measured by participant
Change in smoking | Baseline and every 4 weeks up to month 12
  Test Fagerstrom questionnaire. 6-items. Four items are a yes/no questions rated from 0 to 1; and the two remaining were multiple-choice questions rated from 0 to 3 on a 4-point Likert-type scale.
Change in alcohol use | Baseline and every 4 weeks up to month 12
  Alcohol Use Disorders Identification Test (AUDIT) questionnaire. 10-items, 4-point Likert-scale rated from 0 to 3. A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Change in diet | Baseline and every 4 weeks up to month 12
  14-item Mediterranean diet adherence questionnaire. Each item can be assigned a score of 0 (no adherence to Mediterranean diet) or 1 (adherence). A score of ≤5 is considered low adherence, a score between 6 and 9 is medium adherence, and a score of ≥10 is high adherence.
Change in sleep | Continuously across a 12-month time period
  EmbracePlus wearable device
Change in physiological stress response | Continuously across a 12-month time period
  EmbracePlus wearable device
Change in medication use | Baseline and every day up to month 12
  Non-validated daily medication use questionnaire. 3-items
Adverse side effects | Baseline and every week up to month 12
  Canadian ADHD Resource Alliance. CADDRA Patient ADHD Medication Form. 5-item questionnaires. 3-items record changes in ADHD symptom control, side effects and quality of life using a 7-item Likert-scale, rated from -3 (worse) to 3 (better). 1 item records global changes using a 5-item Likert-scale, rated from 0 (marked deterioration) to 3 (mark improvement). 1 item lists all common side effects of ADHD medication, each side effect is rated from 0 (not at all) to 3 (all the time).

CONTACTS AND LOCATIONS:
Overall Officials: Jonna Kuntsi, BSc, MSc, PhD, Principal Investigator — Social, Genetic and Developmental Psychiatry Centre, Institute of Psychiatry, Psychology and Neuroscience, King's College London
Locations (2):
- Vall d'Hebron Research Institute, Barcelona, Spain
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No